CLINICAL TRIAL: NCT05186974
Title: An Open-label, Multicenter, Phase 2 Study of Sacituzumab Govitecan Combinations in First-line Treatment of Patients With Advanced or Metastatic Non-Small-Cell Lung Cancer (NSCLC) Without Actionable Genomic Alterations
Brief Title: Study of Sacituzumab Govitecan Combinations in First-line Treatment of Participants With Advanced or Metastatic Non-Small-Cell Lung Cancer (NSCLC)
Acronym: EVOKE-02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-576-6220; 2021-004280-27 (EudraCT Number); KEYNOTE-D15 (Other: Merck Sharp & Dohme LLC); MK-3475-D15 (Other: Merck & Co., Inc.); 2024-513225-23 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2021-12-23; First posted 2022-01-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sacituzumab govitecan; pembrolizumab; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Sacituzumab Govitecan-hziy (SG) + Pembrolizumab (Cohort A) (Experimental): Participants assigned to Cohorts A according to tumor proportion score (TPS) status will receive SG 10 mg/kg on Days 1 and 8 of a 21-day cycle + pembrolizumab 200 mg on Day 1 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG); Drug: Pembrolizumab
- SG + Pembrolizumab (Cohort B) (Experimental): Participants assigned to Cohorts B according to TPS status will receive SG 10 mg/kg on Days 1 and 8 of a 21-day cycle + pembrolizumab 200 mg on Day 1 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG); Drug: Pembrolizumab
- SG + Pembrolizumab + Carboplatin Safety Run-in (Experimental): Participants will receive SG (de-escalating dose levels: 10.0 mg/kg, 7.5 mg/kg, or 5.0 mg/kg) on Days 1 and 8 of a 21-day cycle + pembrolizumab 200 mg on Day 1 of a 21-day cycle + carboplatin area under the concentration versus time curve (AUC)5 on Day 1 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG); Drug: Pembrolizumab; Drug: Carboplatin
- SG + Pembrolizumab + Cisplatin Safety Run-in (Optional) (Experimental): Participants will receive SG (either 10 mg/kg or 7.5 mg/kg) on Days 1 and 8 of a 21-day cycle + pembrolizumab 200 mg on Day 1 of a 21-day cycle + cisplatin 75 mg/m^2 on Day 1 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG); Drug: Pembrolizumab; Drug: Cisplatin
- SG + Pembrolizumab + Carboplatin or Cisplatin (Cohort C) (Experimental): Participants assigned to Cohort C according to disease status will receive SG RP2D as determined during the safety run-in cohorts on Days 1 and 8 of a 21-day cycle + pembrolizumab 200 mg on Day 1 of a 21-day cycle + carboplatin AUC5 or cisplatin 75 mg/m^2 as determined during the safety run-in cohorts on Day 1 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG); Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin
- SG + Pembrolizumab + Carboplatin or Cisplatin (Cohort D) (Experimental): Participants assigned to Cohort D according to disease status will receive SG RP2D as determined during the safety run-in cohorts on Days 1 and 8 of a 21-day cycle + pembrolizumab 200 mg on Day 1 of a 21-day cycle + carboplatin AUC5 or cisplatin 75 mg/m^2 as determined during the safety run-in cohorts on Day 1 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG); Drug: Pembrolizumab; Drug: Carboplatin; Drug: Cisplatin
- SG + Pembrolizumab + Cisplatin (Cohort E) (Experimental): Participants assigned to Cohort E will receive SG RP2D, as determined following safety review of Cohorts C and D, on Days 1 and 8 of a 21-day cycle + pembrolizumab 200 mg on Day 1 of a 21-day cycle + cisplatin 75 mg/ m^2 on Day 1 of a 21-day cycle.
  Interventions: Drug: Sacituzumab Govitecan-hziy (SG); Drug: Pembrolizumab; Drug: Cisplatin

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy (SG) — Administered intravenously
  Other Names: GS-0132; IMMU-132
Drug: Pembrolizumab — Administered intravenously
  Other Names: KEYTRUDA®
Drug: Carboplatin — Administered intravenously
  Other Names: Paraplatin®
  Arms: SG + Pembrolizumab + Carboplatin Safety Run-in; SG + Pembrolizumab + Carboplatin or Cisplatin (Cohort C); SG + Pembrolizumab + Carboplatin or Cisplatin (Cohort D)
Drug: Cisplatin — Administered intravenously
  Other Names: Platinol®
  Arms: SG + Pembrolizumab + Carboplatin or Cisplatin (Cohort C); SG + Pembrolizumab + Carboplatin or Cisplatin (Cohort D); SG + Pembrolizumab + Cisplatin (Cohort E); SG + Pembrolizumab + Cisplatin Safety Run-in (Optional)

SUMMARY:
The goal of this clinical study is to learn more about the study drug, sacituzumab govitecan-hziy (SG), and its dosing in combination with pembrolizumab or pembrolizumab and a platinum agent (carboplatin or cisplatin), in participants with advanced or metastatic (cancer that has spread) non-small-cell lung cancer (NSCLC).

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals with pathologically documented evidence of Stage IV non-small cell lung Cancer (NSCLC) disease at the time of enrollment
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) as per RECIST Version 1.1 criteria by investigator
* No prior systemic treatment for metastatic NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Adequate hematologic counts
* Adequate hepatic function

Key Exclusion Criteria:

* Mixed SCLC and NSCLC histology
* Active second malignancy
* NSCLC that is eligible for definitive local therapy alone
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has had an allogenic tissue/solid organ transplant.
* Has severe (≥ Grade 3) hypersensitivity to SG, pembrolizumab, carboplatin, or cisplatin, their metabolites, or formulation excipient
* Has received radiation therapy to the lung
* Individuals may not have received systemic anticancer treatment within the previous 6 months
* Is currently participating in or has participated in a study of an investigational agent
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Known active central nervous system (CNS) metastases
* History of cardiac disease
* Active chronic inflammatory bowel disease
* Active serious infection requiring antibiotics
* Active or chronic hepatitis B infection
* Positive hepatitis C antibody
* Positive serum pregnancy test or women who are lactating

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate as Assessed by Independent Review Committee (IRC) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to 22 Months
Percentage of Participants Experiencing Dose-limiting Toxicities (DLTs) per Dose Level in the Safety Run-in Cohorts | First dose date up to 21 days

SECONDARY OUTCOMES:
Progression-free Survival as Assessed by IRC per RECIST Version 1.1 | Up to 24 Months
Overall Survival | Up to 24 Months
Duration of Response as Assessed by IRC per RECIST Version 1.1 | Up to 24 Months
Disease Control Rate as Assessed by IRC per RECIST Version 1.1 | Up to 24 Months
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 24 Months plus 30 days
Percentage of Participants Experiencing Clinical Laboratory Abnormalities | First dose date up to 24 Months plus 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (101):
- United States (22):
  - Alaska Oncology and Hematology, LLC., Anchorage, Alaska
  - Beverly Hills Cancer Center, Beverly Hills, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology/Oncology - Santa Monica, Los Angeles, California
  - UC Irvine Health, Orange, California
  - Stanford Cancer Institute, Stanford, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital Central Research Department, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Orchard Healthcare Research Inc., Skokie, Illinois
  - Kansas City Veterans Affairs Medical Center, Westwood, Kansas
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Weill Cornell Medical/New York-Presbyterian Hospital, New York, New York
  - Great Lakes Cancer Care, Williamsville, New York
  - Wake Forest Baptist Health - High Point Medical Center, High Point, North Carolina
  - FirstHealth Outpatient Cancer Center, Pinehurst, North Carolina
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - OSU Brain & Spine Hospital, Columbus, Ohio
  - Siouxland Regional Cancer Center dba June E. Nylen Cancer Center, North Sioux City, South Dakota
- Australia (10):
  - Southern Highlands Cancer Centre, Bowral, New South Wales
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - St George Private Hospital, Kogarah, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Ashford Cancer Centre Research, Windsor Gardens, South Australia
  - Peninsula Health - Frankston Hospital, Frankston, Victoria
  - Western Health - Sunshine Hospital, Melbourne, Victoria
  - Joondalup Health Campus, Joondalup, Western Australia
- Canada (2):
  - CIUSSS Saguenay Lac St-Jean, Québec
  - McGill University Health Centre, Québec
- France (11):
  - APHP - Hôpital Ambroise Paré, Boulogne-Billancourt
  - CHRU de Brest - Hopital Morvan, Brest
  - Centre Francois Baclesse, Caen
  - CHU de CAEN, Caen
  - Centre Jean Perrin - 58 rue Montalembert, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Institut Curie, Paris
  - CHU de Bordeaux Hopital Haut leveque, Pessac
  - Hospices Civils de Lyon, Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
- Germany (9):
  - Evangelische Lungenklinik Berlin Krakenhausbetriebs GmBH, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitatsklinikum Koln, Klinik I fur Innere Medizin, Cologne
  - Klinikum Esslingen GmbH, Klinik fur Kardiologie, Angiologie und Pneumologie, Esslingen am Neckar
  - Universitatsklinikum Frankfurt, Frankfurt
  - Asklepios Fachkliniken Munchen-Gauting, Zentrum fur Pneumologie und Thoraxchirugie, Gauting
  - LungenClinic Grosshansdorf, Großhansdorf
  - Martha-Maria Krankenhaus Halle Dölau gGmbH, Halle
  - LKI Lungenfachklinik Immenhausen, Immenhausen
- Hong Kong (4):
  - Department of Clinical Oncology, The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Hong Kong United Oncology Center, Kowloon
- Italy (5):
  - ASST Spedali Civili di Brescia, Brescia
  - AOU Policlinico Vittorio Emanuele - POG Rodolico, Catania
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - IRCCS Istituti Fisioterapicic Ospitalieri - Istituto Nazionale Tumori Regina Elena, Rome
  - IRCCS Instituto Clinico Humanitas, Rozzano
- Malaysia (7):
  - Sultan Ismail Hospital, Johor Bahru
  - Hospital Raja Perempuan Zainab II, Kota Bharu
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Sarawak General Hospital, Kuching
  - Institut Kanser Negara, Putrajaya
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si
  - Gachon University Gil Medical Center, Inchon
  - Asan Medical Center, Seoul
  - Seoul Metropolitan Government - Seoul National University Boramae Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (13):
  - Complejo Hospitalario Universitario A Coruna. Hospital Teresa Herrera, A Coruña
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Duran i Reynals, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Puerta de Hierro de Majadahonda, Majadahonda
  - Clinica Universidad de Navarra - Pamplona, Pamplona
  - Hospital Regional Universitario de Malaga-Hospital Civil, Rincón de la Victoria
  - Complejo Hospitalario Universitario de Santiago de Compostela CHUS_Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-DA Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chi Mei Hospital - Liouying, Liouying Dist.
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, Taipei
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital (CGMH), Taoyuan
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Guy's and St Thomas' NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-576-6220